CLINICAL TRIAL: NCT03531996
Title: The Longitudinal Evaluation of Autoimmune Pulmonary Alveolar Proteinosis
Acronym: LongPAP
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2017-7514; U54HL127672 (NIH)
Record Dates: First submitted 2018-05-07; First posted 2018-05-22 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Autoimmune Pulmonary Alveolar Proteinosis
Keywords: Pulmonary Surfactant; Rare Lung Disease; Registry
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis, Acquired

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Biospecimens retained will be serum, plasma, and DNA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The major goal of this study is to conduct a prospective, longitudinal study of autoimmune PAP to examine outcome measures for disease severity of potential use in clinical practice and/or clinical research studies. These results will impact the field by: 1) improving an understanding of the clinical course of autoimmune PAP, 2) providing information on various clinical outcome and quality of life outcome measures to guide patients and physicians in making treatment choices, and 3) facilitate the development of pharmaco-therapeutics for autoimmune PAP and 4) better informing PAP researchers.

DETAILED DESCRIPTION:
PAP is a rare syndrome of surfactant accumulation and resulting hypoxemic respiratory failure that occurs in a number of diseases classified pathogenically into three groups: primary PAP (caused by disruption of GM-CSF signaling - autoimmune PAP, hereditary PAP), secondary PAP (caused by reduction in alveolar macrophage numbers and/or functions), and surfactant dysfunction-related PAP (caused by mutations in genes required for normal surfactant production). In current clinical practice, PAP is diagnosed based on a lung biopsy; an approach that is not able to identify the PAP-causing disease in anyone. Current therapy involves the physical removal of surfactant by a procedure in which the lungs are repeatedly filled with saline and emptied - whole lung lavage, which is invasive, inefficient, and not widely available, especially for children. Importantly, research advances have elucidated the pathogenesis of diseases causing PAP in most patients and have identified new diagnostic and therapeutic approaches. Simple blood-based research tests can now identify the PAP-causing disease in about 95% of patients. Further, several promising potential disease-specific therapies are currently in development. The long-term goals of the Rare Lung Diseases Consortium include improving the diagnosis and therapy of people with PAP. A major goal of this protocol is to conduct a prospective, longitudinal study of autoimmune PAP to examine outcome measures for disease severity for potential use in clinical practice and/or clinical research studies. The investigator's central hypothesis is that a prospective, longitudinal study of autoimmune PAP patients will facilitate the identification of useful outcome measures for use in clinical practice and/or clinical research studies. The specific objectives of the study are to: 1) evaluate blood-based biomarkers of PAP lung disease over time in autoimmune PAP patients, 2) evaluate the natural history/clinical course of autoimmune PAP over time, 3) evaluate quality of life measures over time in autoimmune PAP patients, 4) evaluate physiologic measures of disease over time in autoimmune PAP patients, and 5) evaluate radiologic measures of lung disease progression over time in autoimmune PAP patients. The study design will be observational and will involve recruitment, screening, and enrollment of eligible participants and annual collection of clinical data. The experimental approach will be to assess the rate of change in GM-CSF signaling assay parameters from baseline to 24 months. GM-CSF signaling assay parameters include GM-CSF autoantibody (GMAb) level, pSTAT5-Max, STAT5-phosphorylation index (STAT5-PI), GM-CSF signaling index (GM-SI), and GM-CSF EC50. The study will also assess the progression of autoimmune PAP, including but not limited to use of treatment options, the number and types of infections and other inter-current medical issues with quality of life measures, exercise tolerance, and radiologic imaging. Experimental outcomes will evaluate SP-D, cholestenoic acid, and lipid levels. Anticipated results will establish a natural history/clinical course of autoimmune PAP to better serve patients and providers, to better inform PAP researchers, and validate outcome measures and biomarkers for use in future clinical studies of PAP. These results will impact the field by: 1) improving an understanding of the clinical course of autoimmune PAP, 2) providing information on various clinical outcome and quality of life outcome measures to guide patients and physicians in making treatment choices, and 3) facilitate the development of pharmacotherapeutics for autoimmune PAP and 4) better informing PAP researchers.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be provided by:

  * Participant if at least 18 years old -OR-
  * Parent/legal guardian if participant is less than 18 years old -AND-
  * Participant provides assent when appropriate
* History of diagnosis of autoimmune as indicated by a:

  * History of chest CT or x-ray findings compatible with PAP -AND-
  * History of a Positive (Abnormal) serum GMAb test

Exclusion Criteria:

* Individuals who have a serious medical illness that, in the opinion of the investigator, is likely to interfere with completion of the study will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Pulmonary Alveolar Proteinosis
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Longitudinal evaluation of GM-CSF autoantibody levels | Baseline, 1 year, and 2 years
  Change in GM-CSF autoantibody levels in autoimmune PAP patients over time
Longitudinal evaluation of the maximal phospho-STAT5 level after GM-CSF stimulation | Baseline, 1 year, and 2 years
  Change in phospho-STAT5 levels in autoimmune PAP patients over time
Longitudinal evaluation of the STAT5 Phosphorylation Index | Baseline, 1 year, and 2 years
  Change in the STAT5 phosphorylation index in autoimmune PAP patients over time
Longitudinal evaluation of the GM-CSF Signaling Index | Baseline, 1 year, and 2 years
  Change in GM-CSF signaling index in autoimmune PAP patients over time
Longitudinal evaluation of the dose GM-CSF to stimulation 1/2 maximal STAT5 phosphorylation (EC50) | Baseline, 1 year, and 2 years
  Change in GM-CSF EC50 level in autoimmune PAP patients over time

SECONDARY OUTCOMES:
Frequency of therapeutic intervention | Baseline, 1 year, and 2 years
  Change over time in the patient's history of a need for therapeutic intervention
Concurrent infections | Baseline, 1 year, and 2 years
  Change over time in the patient's history of concurrent infections
Blood SP-D | Baseline, 1 year, and 2 years
  Change over time in serum SP-D levels
Blood cholestenoic acid | Baseline, 1 year, and 2 years
  Change over time in cholestenoic acid levels
Blood lipid levels | Baseline, 1 year, and 2 years
  Change over time in blood lipid levels
Quality of Life measured by St. George Respiratory Questionnaire | Baseline, 1 year, and 2 years
  Change over time in the overall health, daily life, and perceived well-being in patients with obstructive airways disease. The questionnaire is divided into two parts: Part 1: Symptoms component (frequency & severity) with a 1, 3 or 12-month recall (best performance with 3- and 12-month recall); Part 2: Activities that cause or are limited by breathlessness; Impact components (social functioning, psychological disturbances resulting from airways disease) refer to current state as the recall.
Shortness of breath measured by San Diego Dyspnea Score | Baseline, 1 year, and 2 years
  Change over time in the severity of shortness of breath on a 6-point scale (0 = Not at all, 5 = Maximally or unable to do because of breathlessness) during 21 activities of daily living associated with varying levels of exertion. Three additional questions ask about fear of harm from overexertion, limitations, and fear caused by shortness of breath, for a total of 24 items. If patients do not routinely perform an activity, they are asked to estimate their anticipated shortness of breath. A total sum score ranges from 0 to 120.
Minimum SpO2 during a standardized exercise protocol | Baseline, 1 year, and 2 years
  Change over time in the minimum SpO2 during exercise on a scale of 0 to 100. The study will be stopped if the Sp02 reaches 88%.
Time during standardized exercise protocol required for SpO2 to fall below 88% | Baseline, 1 year, and 2 years
  Change over time in the time for the SpO2 to fall below 88% during the standardized exercise protocol while patients step onto and off of a step for 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Trapnell, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trapnell BC, Whitsett JA, Nakata K. Pulmonary alveolar proteinosis. N Engl J Med. 2003 Dec 25;349(26):2527-39. doi: 10.1056/NEJMra023226. No abstract available. PMID 14695413
- [Background] Carey B, Trapnell BC. The molecular basis of pulmonary alveolar proteinosis. Clin Immunol. 2010 May;135(2):223-35. doi: 10.1016/j.clim.2010.02.017. Epub 2010 Mar 25. PMID 20338813
- [Background] Uchida K, Nakata K, Carey B, Chalk C, Suzuki T, Sakagami T, Koch DE, Stevens C, Inoue Y, Yamada Y, Trapnell BC. Standardized serum GM-CSF autoantibody testing for the routine clinical diagnosis of autoimmune pulmonary alveolar proteinosis. J Immunol Methods. 2014 Jan 15;402(1-2):57-70. doi: 10.1016/j.jim.2013.11.011. Epub 2013 Nov 23. PMID 24275678